CLINICAL TRIAL: NCT04935580
Title: Frontline Therapy of GC012F Injection in Transplant Eligible Newly Diagnosed Multiple Myeloma Patients With High-Risk Profile
Brief Title: Study of FasT CAR-T GC012F Injection in High Risk TE NDMM Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Collaborators: Gracell Biotechnologies (Shanghai) Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Juan Du, Director of Hematology Department, Shanghai Changzheng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC012F-32
Record Dates: First submitted 2021-06-13; First posted 2021-06-23 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GC012F treatment (Experimental): GC012F will be infused at a dose of1- 3 x 10^5 CAR+ T cells/kg after receiving lymphodepleting chemotherapy. Lenalidomide maintenance therapy will be given post month 6 at physicians' choice.
  Interventions: Biological: GC012F injection

INTERVENTIONS:
Biological: GC012F injection — GC012F injection is an autologous dual CAR-T targeted BCMA and CD19. A single infusion of CAR-T cells will be administered intravenously.

SUMMARY:
This is a single-arm, single-center, open-label clinical study to evaluate the safety and efficacy of GC012F in high-risk, transplant eligible patients with NDMM.

DETAILED DESCRIPTION:
Twenty evaluable subjects are planned to be enrolled in this study. Apheresis will be carried out in subjects who meet eligible criteria, and total 2 cycles of induction therapy (three-drug combination regimen based on bortezomib with details determined by the investigator according to the patient's condition) will be selectively given to subjects before or after apheresis. Next, subjects will receive a single infusion of GC012F, and the efficacy assessments will be performed at 1 month, 3 months, and every 3 months within 2 years until the end of the trial (MRD testing is required for each efficacy assessment),

1.Efficacy assessments performed at the 1st and 3rd months after infusion:

1. <PR: Protocol change or transplantation or follow-up decided by the investigator.
2. ≥PR: MRD positive: Protocol change or transplantation or follow-up decided by the investigator.

MRD negative: Wait for next follow-up.

2.Efficacy assessments performed at the 6th month after infusion and every 3 months thereafter:

1. MRD positive: Protocol change or transplantation or follow-up decided by the investigator.
2. MRD negative: Whether to carry out maintenance treatment using lenalidomide until the end of the trial will be determined by the investigator.

After signing the informed consent form (ICF), subjects will be followed up for efficacy and safety until 2 years after GC012F infusion, or disease progression, or death, or withdrawal of consent, or any intolerable toxicity, whichever comes first. All AEs in subjects, especially infection related symptoms and signs, will be closely monitored during follow-up, and prophylactic treatment will be administered according to clinical practice when necessary. In case of disease progression within 2 years after GC012F infusion, treatment will be administered according to clinical practice, and the survival follow-up (only for the survival status) will be performed every 12 weeks±14 days (2 weeks) until 2 years after infusion, or death, or withdrawal of consent, whichever comes first. For subjects who have undergone transportation or any other clinical routine treatments after GC012F infusion, survival follow-up will be also performed as described above.

ELIGIBILITY:
Inclusion Criteria:

* Patients should meet all of the following criteria:

  1. ≥18 years of age at the time of signing informed consent-upper age limit 70;
  2. High-risk defined as meet one or more of the following criteria at screen:

     1. R-ISS stage II or III;
     2. LDH > the upper limit of normal;
     3. Meet one or more of cytogenetic high risk defined by: del 17p, t(4:14), t(14:16); Gain 1q21≥ 4 copies;
     4. Patients with extramedullary disease;
     5. IgD or IgE subtype;
     6. Meet one or more high-risk definition of mSMART3.0;
  3. Documented evidence of multiple myeloma at diagnosis as defined by IMWG guidelines CRAB (calcium elevation, renal insufficiency, anemia, and bone abnormalities)/SLiM criteria, monoclonal plasma cells in the bone marrow ≥10% or presence of a biopsy proven plasmacytomas, and measurable secretory disease according to IMWG criteria meet one or more of the following criteria at screening:

     1. Serum M protein ≥ 1 g/dL;
     2. Urine M protein ≥ 200 mg/24h;
     3. Serum free light chain sFLC ≥ 10 mg/dL with abnormal serum immunoglobulin κ/λ free light chain ratio.
  4. ECOG score was 0-2 at screen;
  5. Estimated life expectancy ≥3 months;
  6. Absolute neutrophil count (ANC) ≥ 1.5×10^9/L without use of growth factors;
  7. Platelet count ≥ 75×10^9/L without transfusion support within 7 days before the screen;
  8. Hemoglobin≥ 80 g/L;
  9. Adequate functional reserve of organs:

     1. ALT/AST ≤ 2.5× UNL (upper normal limit);
     2. Creatinine clearance ≥ 40mL/min, or serum creatinine level ≤177μmol/L，may be calculated or measured according to local practice;
     3. Serum total bilirubin ≤ 1.5× UNL, except in subjects with congenital bilirubinemia, such as Gilbert syndrome, then direct bilirubin ≤ 1.5× UNL;
     4. The left ventricular ejection fraction (LVEF)≥50%, and no clinically significant ecg abnormalities were found;
     5. Basic oxygen saturation in natural indoor air: SPO2>92%.
  10. Adequate venous access for apheresis collection, and no other contraindications to apheresis;
  11. Subjects and sexual partner with fertility are willing to use effective and reliable method of contraception for at least 1 year after CART cell infusion, serum HCG should be negative in females with fertility both at screening andbaseline;
  12. Subjects must sign a written informed consent.

Exclusion Criteria:

* Patients should be excluded if they meet any one of the following criteria:

  1. Patients with purely non-secretory MM;
  2. Subject has had radiation therapy within 14 days of screening;
  3. Subjects has plasma cell leukemia or POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes);
  4. Subjects has a diagnosis of primary amyloidosis, Waldenstroem's disease, monoclonal gammopathy of undetermined significance, or smoldering multiple myeloma;
  5. Having other tumors (excluding non-melanoma skin cancer and cervical cancer in situ bladder cancer and breast cancer that have been disease-free for more than 5 years);
  6. Overt clinical evidence of dementia or altered mental status; any history of central nervous system (CNS) disease or neurodegenerative disorder, such as epilepsy, seizures, paralysis, aphasia, stroke, severe brain damage, dementia, Parkinson's disease, psychosis;
  7. History of hereditary diseases such as Fanconi anemia, Schrader syndrome, Costerman syndrome, or any other known bone marrow failure syndrome;
  8. Clinically significant cardiac disease including: uncontrolled cardiac arrhythmia or clinically significant ECG abnormalities, grade III-IV heart failure or myocardial infarction cardiac angioplasty or stenting unstable angina or other clinically significant cardiac conditions within one year prior to enrollment;
  9. Presence of any indwelling catheter or drainage tube (e.g., percutaneous nephrostomy catheter indwelling catheter bile drainage tube or pleural/peritoneal/pericardial catheter) permits the use of a dedicated central venous catheter;
  10. Subjects is exhibiting clinical signs of meningeal involvement of multiple myeloma;
  11. A positive virological result for any of the following: HIV, HCV, HBsAg, TPPA;
  12. Other severe viral or bacterial infections or uncontrolled systemic fungal infections are present;
  13. Subjects with a history of severe hypersensitivity;
  14. There is a history of an autoimmune disease (e.g., Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus) that has resulted in terminal organ damage or requires systemic immunosuppressive/disease modulating drugs in the past 2 years;
  15. Presence of lung disease (such as pulmonary fibrosis);
  16. Subjects has had major surgery within 2 weeks before screen or has not fully recovered from surgery, or has surgery planned during the time the subject is expected to participate in the study;
  17. Poor compliance due to factors such as physiological family, social geography, etc., and inability to comply with the research program and follow-up plan;
  18. Pregnant or lactating women, or men who are planned to have babies during the period of participation in the study or within 1 year of receiving treatment;
  19. Investigator assessment deemed to be ineligible.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-06-28 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AE) after GC012F infusion | Up to 1 year after patients infused with GC012F injection
  An assessment of severity grade will be made according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), with the exception of cytokine release syndrome (CRS), and immune effector cell-associated neurotoxicity syndrome (ICANS). CRS and ICANS should be evaluated according to the American Society for Transplantation and Cellular Therapy (ASTCT) consensus grading
Overall response rate (ORR) as measured by International Myeloma Working Group (IMWG) criteria after GC012F infusion | Up to 2 years after patients infused with GC012F injection
  ORR defined as proportion of patients achieving PR or better based on IMWG defined response criteria
Percentage of patients with minimal residual disease (MRD) negative(tested by NGF at sensitivity of 10e-5 to 10e-4) at landmark analysis of 1/3/6/12/18/24 months post GC012F infusion | Up to 2 years after patients infused with GC012F injection
  MRD negative rate is defined as the proportion of participants who achieve MRD negative status by the respective time point
Progress free survival (PFS) at 6 months, 12 months and 24 months after GC012F infusion | Up to 2 years after patients infused with GC012F injection
  PFS defined as time from date of GC012F infusion to date of first documented disease progression, or death due to any cause, whichever occurs first. DOR defined as time form Month 1 after GC012F infusion to date of 1st documented PD if patients' response deeper or keeping sCR after CAR-T infusion.
Duration of response (DOR) at 6 months, 12 months and 24 months after GC012F infusion | Up to 2 years after patients infused with GC012F injection
  DOR defined as time form Month 1 after GC012F infusion to date of 1st documented PD if patients' response deeper or keeping sCR after CAR-T infusion.

SECONDARY OUTCOMES:
Overall survival (OS) after GC012F infusion | Up to 2 years after patients infused with GC012F injection
  Response is defined as participant has met all criteria for PR or better according to IMWG criteria
Time to first response (TTR) after GC012F infusion | Up to 2 years after patients infused with GC012F injection
  Response is defined as participant has met all criteria for PR or better according to IMWG criteria
Time to best response (TBR) after GC012F infusion | Up to 2 years after patients infused with GC012F injection
  Response is defined as participant has met all criteria for PR or better according to IMWG criteria
Change from Baseline in Health-related Quality of Life (HRQoL) as Measured by EORTC QLQ-C30 | Baseline up to study completion ( 2 years after GC012F Infusion on Day 0
  HRQoL will be assessed by the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core-30 (QLQC30) items. Subscale and single item scores are reported on a 0-100 scale with higher scores representing better global health status, better functioning, and worst symptoms.
Change from Baseline in HRQoL as Measured by EORTC QLQ-MY20 | Baseline up to study completion ( 2 years after GC012F Infusion on Day 0
  HRQoL will be assessed by the EORTC QLQ-Multiple Myeloma ((MY20) module items. Subscale and single item scores are reported on a 0-100 scale with higher scores representing better global health status, better functioning, and worst symptoms.
Change from Baseline in Participant-reported Health Status Measured by EQ-5D- 5L | Baseline up to study completion ( 2 years after GC012F Infusion on Day 0
  Participant-reported health status measured by the EuroQol Group 5-dimension, 5-level (EQ-5D-5L) questionnaire. A total utility score is reported based on the health status, ranging from 0 to 1, where higher values indicate better health utility. The visual analog scale ranges from 0 to 100 where higher values indicate better overall health status.
Change from Baseline in Pain Measured by PGIS Scale [Time Frame: Baseline up to study completion | Baseline up to study completion ( 2 years after GC012F Infusion on Day 0
  Participant reported pain measured by Patient Global Impression of Severity (PGIS) Scale. The PGIS is a single item to assess pain severity. The 5-point verbal rating scale ranged from 1 (none) to 5 (very severe).
Level of CAR-T Cell Expansion (proliferation), and Persistence | Up to 2 years after patients infused with GC012F injection
  Levels of GC012F cell expansion (proliferation), and persistence via monitoring CAR-T positive cell counts and CAR transgene level will be reported.
Cytokines in the peripheral blood after GC012F infusion | Up to 2 years after patients infused with GC012F injection
  Serum concentrations of Granulocyte-macrophage Colony Stimulating Factor (GM-CSF), interleukin (IL)-6, IL-10, interferon-gamma (IFN-γ), soluble BCMA (sBCMA) and TNF-α after GC012F infusion
Serum concentrations of C-reaction protein (CRP) | Up to 2 years after patients infused with GC012F injection
  Serum concentrations of C-reaction protein (CRP)
Number of patients with Anti-GC012F Antibodies, replication-competent lentivirus (RCL) after GC012F infusion | Up to 2 years after patients infused with GC012F injection
  Number of patients exhibiting anti-drug antibodies for GC012F and RCL will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Juan Du, MD, Principal Investigator — Shanghai Changzheng Hospital
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China